CLINICAL TRIAL: NCT01099098
Title: Prevalence of Latent Tuberculosis (TB) Infection Diagnosed by Interferon-gamma Release Assay and Tuberculin Skin Tests in Patients With Old Healed TB
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Joon Yim / Associate Professor, Seoul National University Hospital
Other Study IDs: H-0909-054-295
Record Dates: First submitted 2010-04-04; First posted 2010-04-06 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Tuberculosis
Keywords: People who have fibrosis or nodules in their upper lobe of the lung
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with TB sequelae
- People without TB sequelae

SUMMARY:
We easily regard nodules and fibrosis in upper lobes of lung as TB sequelae. The aim of this study is to confirm the prevalence of latent TB infection diagnosed by interferon-gamma release assay and tuberculin skin tests in patients with old healed TB.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* Patients with TB sequelae in their CXR

Exclusion Criteria:

* Patients on immune-suppressants

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with TB sequelae in their CXR
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of latent TB infection | At enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea